CLINICAL TRIAL: NCT01118585
Title: Prospective Outcome Evaluation of Transoral Incisionless Fundoplication (TIF) for the Treatment of Gastroesophageal Reflux Disease (GERD): The TIF Registry Study
Brief Title: Transoral Incisionless Fundoplication (TIF) Registry Study for Treatment of Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoGastric Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D00960
Record Dates: First submitted 2010-04-30; First posted 2010-05-06 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Gastroesophageal Reflux Disease; Hiatal Hernia
Keywords: GERD; Esophagitis; Fundoplication; Anti-reflux surgery; PPI dependent
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal; Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TIF Procedure (Other): Intervention: Transoral incisionless fundoplication procedure using the EsophyX device. During general anesthesia the EsophyX device is introduced trans orally into the stomach and used to created a 270 degree, 3cm in length, wrap at the distal end of the esophagus to treat GERD.. .
  Interventions: Procedure: TIF Procedure

INTERVENTIONS:
Procedure: TIF Procedure — The TIF procedure results in the creation of an esophago-gastric fundoplication extending up to 4 cm above the Z-line and 270 degrees around the esophagus.
  Other Names: TIF - Transoral Incisionless fundoplication

SUMMARY:
The study objective is to evaluate the safety and efficacy of TIF among a broad range of GERD patients treated in routine clinical practice at multiple centers across the United States.

DETAILED DESCRIPTION:
Primary Effectiveness Endpoint: Typical and atypical GERD symptom elimination (scores ≤ 2 to each question) or clinically significant improvement (≥ 50% reduction in total scores) at 6-month follow-up compared to baseline.

Secondary Effectiveness Endpoints: GERD symptom elimination or clinically significant improvement at 12-month follow-up, 24-month follow-up and 36-month follow-up; complete discontinuation of PPIs; normalization of esophageal acid exposure; significant reduction in reflux episodes; healing of reflux esophagitis; reduction of hiatal hernia; safety supported by low incidence of serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* GERD for > 1 year
* History of daily PPIs use for > 6 months
* Moderate to severe typical or atypical GERD symptoms off PPIs
* Complete (responders) or partial (nonresponders) symptom control on PPIs
* Deteriorated gastroesophageal junction (Hill grade II or III)
* Proven gastroesophageal reflux by either endoscopy, ambulatory pH or barium swallow testing
* Willingness to undergo pH/impedance testing, if required
* Willingness to cooperate with the postoperative diet for 6 weeks
* Availability for follow up visits at 6 months and 12 months
* Willingly and cognitively signed informed consent

Exclusion Criteria:

* BMI > 35
* Incompletely reducible hiatal hernia with residual of > 5 mm
* Esophagitis grade D
* Barrett's Esophagus > 2 cm
* Esophageal ulcer
* Fixed esophageal stricture or narrowing
* Portal hypertension and/or varices
* Active gastro-duodenal ulcer disease
* Gastric outlet obstruction or stenosis
* Gastroparesis or delayed gastric emptying confirmed by solid-phase gastric emptying study, if patient complains of postprandial satiety during assessment
* Coagulation disorder
* History of any of the following: resective gastric or esophageal surgery, antireflux surgery with anatomy unsuitable for TIF procedure per physician judgment, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum, achalasia, scleroderma or dermatomyositis, eosinophilic esophagitis, or cirrhosis
* Pregnancy or plans of pregnancy in the next 12 months
* Enrollment in another device or drug study that may confound the results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2010-05; Primary Completion 2015-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Gastroesophageal Reflux Disease (GERD) symptom elimination | 6-month follow-up
  GERD symptoms (typical and atypical) will be evaluated using three disease-specific standardized questionnaires: GERD-HRQL (Health-related Quality of Life), GSRS (GERD Symptom Rating Score), and RSI (Reflux Symptom Index).

SECONDARY OUTCOMES:
Elimination of Proton Pump Inhibitor (PPI) usage | at 12-, 24- and 36-month follow-up
  Elimination of Proton Pump Inhibitor (PPI) usage
Esophageal acid exposure | at 6-, 12-, 24- and 36-month follow-up
  Normalization of esophageal acid exposure is defined as ≤ 4.3% of 24-hour period or ≤ 5.3% of 48-hour period at pH < 4.
Healing of reflux esophagitis | at 12, 24- and 36-month follow-up
  Healing of reflux esophagitis
Safety outcomes | first 30 days
  Incidence of anticipated and unanticipated adverse events
Long-term Gastroesophageal Reflux Disease (GERD) symptom elimination | at 12-, 24- and 36-month follow-up
  GERD symptom elimination based on GERD-HRQL, GSRS and RSI scores.

CONTACTS AND LOCATIONS:
Overall Officials: Reginald CW Bell, MD, FACS, Principal Investigator — SurgOne P.C.
Locations (14):
- United States (14):
  - Mt. Graham Regional Medical Center, Safford, Arizona
  - Tempe St. Luke's Hospital, Tempe, Arizona
  - Swedish Medical Center and SurgOne P.C., Englewood, Colorado
  - Munroe Regional Hospital, Ocala, Florida
  - St Mary's Hospital, Hobart, Indiana
  - Livingston Hospital and Healthcare Services, Inc. CAH, Salem, Kentucky
  - The Surgeons Group of Baton Rouge, Baton Rouge, Louisiana
  - Allegan Surgical Associates, Allegan, Michigan
  - Crossville Medical Group, Crossville, Tennessee
  - Ihde Surgical Group, PA, Arlington, Texas
  - The University of Texas Health Science Center, Houston, Texas
  - Master Center for Minimally Invasive Surgery, Southlake, Texas
  - Utah County Surgical Associates, Provo, Utah
  - Reston Hospital, Reston, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Click here for more information about this study: TIF Registry study — http://www.endogastricsolutions.com